CLINICAL TRIAL: NCT03236558
Title: Thymic Generation of Regulatory T Lymphocytes in Type I Diabetes Patients.
Brief Title: The Role of the Thymus in Type I Diabetes.
Acronym: TregDiab
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of Financial support
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/16/8254
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Type1 Diabetes
Keywords: Type 1 diabetes; Juvenile diabetes; Immune-tolerance; Regulatory T lymphocyte; Treg; TCR; Repertoire
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with diabetes (Experimental): T1D patients with blood collection
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — Ten cc of peripheral blood will be taken from patients and healthy controls as soon as possible after T1D diagnosis of the former.

SUMMARY:
Regulatory T lymphocytes play a major role in the protection from autoimmune pathology. Defects in immunosuppression mediated by these cells is therefore suspected to contribute to these diseases. This issue has very little been studied in humans.Regulatory T cells emigrated from the thymus will be isolated from the blood of patients and healthy controls. The repertoire of antigen-receptors will be analysed by high throughput sequencing and its diversity estimated using appropriate statistical models borrowed from ecology.

DETAILED DESCRIPTION:
In the thymus of an animal model of type I diabetes, the population of regulatory T cells expresses a repertoire of antigen receptors that is approximately ten-fold less diverse than that found in mice resistant to autoimmune pathology. Genetic models later showed that this reduced diversity was involved in the susceptibility to diabetes. Researchers study the diversity of the TCR expressed by regulatory T cells from paediatric type I diabetes patients and controls. Regulatory T cells emigrated from the thymus will be isolated from the blood of patients and healthy controls. The repertoire of antigen-receptors will be analysed by high throughput sequencing and its diversity estimated using appropriate statistical models borrowed from ecology.

ELIGIBILITY:
Inclusion Criteria:

* type I diabetes patient
* having at least one age-matched sibling (healthy control)

Exclusion Criteria:

* other immunopathology
* treatment with any anti-inflammatory or immunosuppressive drugs
* puberty
* legal protection

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Variability of the diversity of antigen-receptors' repertoires, expressed by regulatory T cells from type I diabetes patients and healthy controls. | Day 1
  Treg from the pediatric patients and the control subjects' blood will be isolated by cytometry, the messenger ribonucleic acid (mRNA) of these cells will be isolated, and the analysis of the alpha and beta chains of the TCRs will be carried out by high-throughput sequencing.

SECONDARY OUTCOMES:
Ratio between TCR diversities expressed by Treg cells vs. conventional T cells. | Day 1
  Treg from the pediatric patients and the control subjects' blood will be isolated by cytometry, the mRNA of these cells will be isolated, and the analysis of the alpha and beta chains of the TCRs will be carried out by high-throughput sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Le Tallec, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Background] Ferreira C, Singh Y, Furmanski AL, Wong FS, Garden OA, Dyson J. Non-obese diabetic mice select a low-diversity repertoire of natural regulatory T cells. Proc Natl Acad Sci U S A. 2009 May 19;106(20):8320-5. doi: 10.1073/pnas.0808493106. Epub 2009 Apr 9. PMID 19359477
- [Background] Thiault N, Darrigues J, Adoue V, Gros M, Binet B, Perals C, Leobon B, Fazilleau N, Joffre OP, Robey EA, van Meerwijk JP, Romagnoli P. Peripheral regulatory T lymphocytes recirculating to the thymus suppress the development of their precursors. Nat Immunol. 2015 Jun;16(6):628-34. doi: 10.1038/ni.3150. Epub 2015 May 4. PMID 25939024
- [Background] Steffens CM, Al-Harthi L, Shott S, Yogev R, Landay A. Evaluation of thymopoiesis using T cell receptor excision circles (TRECs): differential correlation between adult and pediatric TRECs and naive phenotypes. Clin Immunol. 2000 Nov;97(2):95-101. doi: 10.1006/clim.2000.4938. PMID 11027449
- [Background] Calder AE, Hince MN, Dudakov JA, Chidgey AP, Boyd RL. Thymic involution: where endocrinology meets immunology. Neuroimmunomodulation. 2011;18(5):281-9. doi: 10.1159/000329496. Epub 2011 Sep 22. PMID 21952680
- [Background] Sakaguchi S, Miyara M, Costantino CM, Hafler DA. FOXP3+ regulatory T cells in the human immune system. Nat Rev Immunol. 2010 Jul;10(7):490-500. doi: 10.1038/nri2785. Epub 2010 Jun 18. PMID 20559327
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396